CLINICAL TRIAL: NCT04186871
Title: A Randomized, Placebo-Controlled, Double-Blind, Multicenter Study to Assess the Efficacy and Safety of Branebrutinib Treatment in Subjects With Active Systemic Lupus Erythematosus or Primary Sjögren's Syndrome, or Branebrutinib Treatment Followed by Open-label Abatacept Treatment in Subjects With Active Rheumatoid Arthritis
Brief Title: Study to Assess Safety and Effectiveness of Branebrutinib Treatment in Participants With Active Systemic Lupus Erythematosus or Primary Sjögren's Syndrome, or Branebrutinib Treatment Followed by Open-label Abatacept Treatment in Study Participants With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM014-029; 2019-002205-22 (EudraCT Number)
Record Dates: First submitted 2019-11-28; First posted 2019-12-05 (Actual); Results first posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Autoimmune Disorder; Rheumatoid Arthritis; Systemic Lupus Erythematosus; Primary Sjögren's Syndrome
MeSH Terms: conditions — Autoimmune Diseases; Arthritis, Rheumatoid; Lupus Erythematosus, Systemic | interventions — branebrutinib; Abatacept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Systemic Lupus Erythematosus (SLE): branebrutinib (Experimental)
  Interventions: Drug: branebrutinib
- SLE: placebo (Placebo Comparator)
  Interventions: Drug: branebrutinib placebo
- Primary Sjögren's Syndrome (pSS): branebrutinib (Experimental)
  Interventions: Drug: branebrutinib
- pSS: placebo (Placebo Comparator)
  Interventions: Drug: branebrutinib placebo
- Rheumatoid Arthritis (RA): branebrutinib followed by abatacept (Experimental)
  Interventions: Drug: branebrutinib; Drug: abatacept
- RA: placebo followed by abatacept (Placebo Comparator)
  Interventions: Drug: abatacept; Drug: branebrutinib placebo

INTERVENTIONS:
Drug: branebrutinib — Specified dose on specified days
  Arms: Primary Sjögren's Syndrome (pSS): branebrutinib; Rheumatoid Arthritis (RA): branebrutinib followed by abatacept; Systemic Lupus Erythematosus (SLE): branebrutinib
Drug: abatacept — Specified dose on specified days
  Arms: RA: placebo followed by abatacept; Rheumatoid Arthritis (RA): branebrutinib followed by abatacept
Drug: branebrutinib placebo — Specified dose on specified days
  Arms: RA: placebo followed by abatacept; SLE: placebo; pSS: placebo

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of treatment with branebrutinib treatment in participants with active systemic Lupus Erythematosus (SLE) or Primary Sjögren's Syndrome (pSS), or branebrutinib treatment followed by open-label abatacept treatment in study participants with active Rheumatoid Arthritis (RA).

ELIGIBILITY:
Inclusion Criteria:

Sub-study for Systemic Lupus Erythematosus (SLE)

* Active SLE as defined by the Systemic Lupus Erythematosus International Collaborating Clinics (SLICC) classification
* Diagnosed with SLE more than 24 weeks before screening visit

Sub-study for primary Sjögren's Syndrome (pSS)

* Moderate to severe pSS, meeting ACR-EULAR classification criteria

Sub-study for active Rheumatoid Arthritis (RA)

* Moderate to severe adult-onset RA
* ACR global functional status class I to III

Women and men must agree to follow instructions for methods of contraception.

Exclusion Criteria:

Sub-study for SLE

* Certain other autoimmune diseases and overlap syndromes

Sub-study for pSS

* Certain other immune-mediated diseases, active fibromyalgia, or other medical conditions

Sub-study for RA

* Diagnosis with juvenile arthritis or idiopathic arthritis before age 16

For all sub-studies:

* History of any significant drug allergy
* Active infection, significant concurrent medical condition, or clinically significant abnormalities

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2022-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (81):
- United States (40):
  - Local Institution - 0019, Phoenix, Arizona
  - Local Institution - 0002, Covina, California
  - Local Institution - 0024, Encino, California
  - Local Institution - 0034, San Diego, California
  - Local Institution - 0032, Upland, California
  - Local Institution, Brandon, Florida
  - Local Institution - 0062, DeBary, Florida
  - Local Institution - 0035, Hialeah, Florida
  - Local Institution, Jacksonville, Florida
  - Local Institution - 0029, Plantation, Florida
  - Local Institution - 0009, Lawrenceville, Georgia
  - Local Institution - 0014, Skokie, Illinois
  - Local Institution, Evansville, Indiana
  - Local Institution - 0005, Monroe, Louisiana
  - Local Institution - 0041, Ann Arbor, Michigan
  - Local Institution - 0082, Grand Blanc, Michigan
  - Local Institution - 0096, St Louis, Missouri
  - Local Institution - 0040, St Louis, Missouri
  - Local Institution - 0056, Lincoln, Nebraska
  - Local Institution - 0007, Las Vegas, Nevada
  - Local Institution, Manhasset, New York
  - Local Institution, New York, New York
  - Local Institution - 0008, Charlotte, North Carolina
  - Local Institution - 0006, Salisbury, North Carolina
  - Local Institution, Minot, North Dakota
  - Local Institution - 0023, Oklahoma City, Oklahoma
  - Local Institution - 0022, Oklahoma City, Oklahoma
  - Local Institution - 0010, Duncansville, Pennsylvania
  - Local Institution - 0045, Orangeburg, South Carolina
  - Local Institution - 0021, Summerville, South Carolina
  - Local Institution - 0079, Jackson, Tennessee
  - Local Institution - 0001, Memphis, Tennessee
  - Local Institution - 0092, Colleyville, Texas
  - Local Institution, Dallas, Texas
  - Local Institution - 0063, Houston, Texas
  - Local Institution - 0016, Mesquite, Texas
  - Local Institution - 0030, Plano, Texas
  - Local Institution - 0031, San Antonio, Texas
  - Local Institution, Waco, Texas
  - Local Institution - 0083, Spokane, Washington
- Argentina (3):
  - Local Institution - 0065, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Local Institution - 0047, San Miguel de Tucum, Tucumán Province
  - Local Institution - 0066, San Juan
- Belgium (2):
  - Local Institution - 0064, Ghent
  - Local Institution - 0069, Leuven
- France (3):
  - Local Institution - 0075, Brest
  - Local Institution - 0070, Marseille
  - Local Institution - 0067, Montpellier
- Germany (5):
  - Local Institution - 0038, Berlin
  - Local Institution - 0037, Cologne
  - Local Institution - 0049, Freiburg im Breisgau
  - Local Institution - 0074, Herne
  - Local Institution - 0051, München
- Mexico (8):
  - Local Institution - 0060, Guadalajara, Jalisco
  - Local Institution - 0042, Guadalajara, Jalisco
  - Local Institution - 0113, Zapopan, Jalisco
  - Local Institution - 0102, Cuernavaca, Morelos
  - Local Institution - 0104, Mérida, Yucatán
  - Local Institution - 0114, San Luis Potosí City
  - Local Institution - 0050, San Luis Potosí City
  - Local Institution - 0059, San Luis Potosí City
- Local Institution - 0004, Groningen, Netherlands
- Poland (11):
  - Local Institution - 0094, Bialystok
  - Local Institution - 0089, Bydgoszcz
  - Local Institution - 0072, Bydgoszcz
  - Local Institution - 0012, Elblag
  - Local Institution - 0073, Elblag
  - Local Institution - 0011, Poznan
  - Local Institution - 0091, Torun
  - Local Institution - 0017, Warsaw
  - Local Institution - 0033, Warsaw
  - Local Institution - 0101, Warsaw
  - Local Institution - 0026, Warsaw
- Spain (5):
  - Local Institution - 0028, A Coru
  - Local Institution - 0036, Barcelona
  - Local Institution - 0025, Málaga
  - Local Institution - 0018, Seville
  - Local Institution - 0061, Valencia
- United Kingdom (3):
  - Local Institution - 0076, Leeds
  - Local Institution - 0058, London
  - Local Institution - 0052, Southampton

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were enrolled concurrently for the RA, SLE, and pSS sub-studies.
Groups:
- SLE- Placebo: Participants with systemic lupus erythematosus (SLE) receive placebo once daily (QD) during a 24-week double-blind placebo-controlled treatment period.
- SLE- Branebrutinib: Participants with systemic lupus erythematosus (SLE) receive branebrutinib 9mg once daily (QD) during a 24-week double-blind placebo-controlled treatment period.
- pSS- Placebo: Participants with primary Sjögren's syndrome (pSS) receive placebo once daily (QD) during a 24-week double-blind placebo-controlled treatment period.
- pSS- Branebrutinib: Participants with primary Sjögren's syndrome (pSS) receive branebrutinib 9mg once daily (QD) during a 24-week double-blind placebo-controlled treatment period.
- RA- Placebo: Participants with rheumatoid arthritis (RA) receive placebo once daily (QD) during a 12-week double-blind placebo-controlled treatment period, followed by an additional 12 weeks of treatment with open-label abatacept.
- RA- Branebrutinib: Participants with rheumatoid arthritis (RA) receive branebrutinib 9mg once daily (QD) during a 12-week double-blind placebo-controlled treatment period, followed by an additional 12 weeks of treatment with open-label abatacept.
Period: Overall Study
Arm/Group | SLE- Placebo | SLE- Branebrutinib | pSS- Placebo | pSS- Branebrutinib | RA- Placebo | RA- Branebrutinib
Started | 5 | 15 | 4 | 10 | 21 | 64
Double Blind Period | 5 | 15 | 4 | 10 | 21 | 64
Open Label Period (The Open Label Period was available to RA sub-study participants only.) | 0 | 0 | 0 | 0 | 20 | 61
Completed | 3 | 11 | 4 | 9 | 20 | 58
Not Completed | 2 | 4 | 0 | 1 | 1 | 6
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0 | 1 | 1
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 0 | 2
Not completed — Study terminated by sponsor | 1 | 2 | 0 | 1 | 0 | 0
Not completed — Other reasons | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SLE- Placebo | SLE- Branebrutinib | pSS- Placebo | pSS- Branebrutinib | RA- Placebo | RA- Branebrutinib | Total
Number analyzed (Participants) | 5 | 15 | 4 | 10 | 21 | 64 | 119
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.6 (10.99) | 44.2 (12.91) | 47.8 (4.19) | 46.6 (9.28) | 46.0 (12.95) | 50.1 (11.62) | 48.2 (11.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 14 | 4 | 7 | 18 | 45 | 93
  Male | 0 | 1 | 0 | 3 | 3 | 19 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 9 | 0 | 1 | 1 | 7 | 21
  Not Hispanic or Latino | 2 | 6 | 4 | 8 | 20 | 57 | 97
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - Non-Japanese: Asian - Non-Japanese | 0 | 0 | 0 | 0 | 0 | 2 | 2
  Asian - Non-Japanese: Black or African American | 1 | 3 | 0 | 0 | 0 | 2 | 6
  Asian - Non-Japanese: White | 2 | 6 | 4 | 9 | 21 | 59 | 101
  Asian - Non-Japanese: Not Reported | 0 | 0 | 0 | 1 | 0 | 1 | 2
  Asian - Non-Japanese: American Indian or Alaska Native | 2 | 6 | 0 | 0 | 0 | 0 | 8

OUTCOME MEASURES:

1. Primary Outcome: The Percent of Participants With mCLASI Response at Week 24 and Corticosteroid (CS) < 10 mg/Day at Week 20 and Week 24 - SLE
Description: mCLASI response is defined as a decrease of ≥ 50% from baseline mCLASI activity score, in participants with a baseline mCLASI activity score ≥ 10, at Week 24. Baseline values are defined as the last nonmissing value prior to the first dose of study treatment.
  To be considered as meeting the second criterion, the CS (prednisone or equivalent) dose had to remain stable and ≤ 10 mg from Week 16 until Week 24.
  The modified CLASI (mCLASI) is defined as the activity portions of CLASI that describe skin erythema and scale/hypertrophy and inflammation of the scalp. The percentage of patients who entered the study with a positive mCLASI activity score (≥ 10) and who achieved a ≥ 50% decrease from baseline at Week 24 is considered to likely represent a clinically meaningful improvement. The scores are calculated by simple addition based on the extent of the symptoms.
  mCLASI: Modified Cutaneous Lupus Erythematosus Disease Area and Severity Index
Time Frame: Week 24
Population: All treated participants with a baseline mCLASI activity score ≥ 10 at Week 24 (Prespecified for participants in the SLE cohort only).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SLE- Placebo | SLE- Branebrutinib
Number analyzed (Participants) | 5 | 15
Percentage of participants | 60.0 [17.1 to 100] | 33.3 [9.5 to 57.2]
Statistical Analysis 1: Comparison: SLE- Placebo vs SLE- Branebrutinib; Test type: Superiority — RESPONSE DIFFERENCE (95% CI) VS PLACEBO; Response Difference = -27.8, 95% CI 2-sided [-77.5 to 21.9]
Statistical Analysis 2: Comparison: SLE- Placebo vs SLE- Branebrutinib; Test type: Superiority — ODDS RATIO (95% CI) VS PLACEBO; p = 0.3117, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.32, 95% CI 2-sided [0.04 to 2.73]

2. Secondary Outcome: Change From Baseline in SLEDAI-2K Score at Week 24 - SLE
Description: The SLEDAI-2K is a global index providing a total score of overall disease activity ranging from 0 to 105, with higher scores representing more active disease. The SLEDAI index includes 24 items divided into 9 organ systems: neurological, musculoskeletal, renal, mucocutaneous, general, heart, respiratory, vascular, and hematological. Each item is scored based on the severity of the symptom or finding, with higher scores indicating more severe disease activity. The weighted scores for each item range from 0 to 8. To calculate the SLEDAI-2K score, the scores for each of the 24 items are added together.
  Baseline values are defined as the last nonmissing value prior to the first dose of study treatment.
Time Frame: Week 24
Population: All Treated Participants with week 24 measurements (Prespecified for participants in the SLE cohort only).
Measure: Mean (Standard Deviation); unit: Change in "score on a scale"
Arm/Group | SLE- Placebo | SLE- Branebrutinib
Number analyzed (Participants) | 4 | 11
Change in "score on a scale" | -7.0 (5.29) | -7.0 (6.54)
Statistical Analysis 1: Comparison: SLE- Placebo vs SLE- Branebrutinib; Test type: Superiority — ADJUSTED MEAN DIFFERENCE VS PLACEBO; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [-2.8 to 4.9]
Statistical Analysis 2: Comparison: SLE- Placebo; Test type: Equivalence — ADJUSTED MEAN DIFFERENCE AT WEEK 24; Mean Difference (Final Values) = -8.3, 95% CI 2-sided [-11.5 to -5.0]
Statistical Analysis 3: Comparison: SLE- Branebrutinib; Test type: Equivalence — ADJUSTED MEAN DIFFERENCE AT WEEK 24; Mean Difference (Final Values) = -7.2, 95% CI 2-sided [-9.3 to -5.2]

3. Secondary Outcome: Percent of Participants With BICLA Response at Week 24 - SLE
Description: BILAG-based composite lupus assessment (BICLA) response is defined as:
  1. At least one gradation of improvement in baseline BILAG scores in all body systems with moderate or severe disease activity at entry
  2. No new BILAG A or more than one new BILAG B scores
  3. No worsening of total SLEDAI score from baseline
  4. No significant deterioration (< 10%) in PGA and
  5. No treatment failure (initiation of nonprotocol treatment).
  BILAG scores: A (severe disease), B (moderate), C (mild), or D (no activity). Baseline values are defined as the last nonmissing value prior to the first dose of study treatment.
Time Frame: Week 24
Population: All Treated Participants (Prespecified for participants in the SLE cohort only).
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | SLE- Placebo | SLE- Branebrutinib
Number analyzed (Participants) | 5 | 15
Percent of participants | 20.0 [0.5 to 71.6] | 33.3 [11.8 to 61.6]
Statistical Analysis 1: Comparison: SLE- Placebo vs SLE- Branebrutinib; Test type: Superiority — RESPONSE DIFFERENCE VS PLACEBO; Response Difference = 16.7, 95% CI 2-sided [-31.8 to 65.2]
Statistical Analysis 2: Comparison: SLE- Placebo vs SLE- Branebrutinib; Test type: Superiority — ODDS RATIO VS PLACEBO; Odds Ratio (OR) = 2.00, 95% CI 2-sided [0.22 to 18.04]

4. Primary Outcome: The Percent of Participants With Composite Response at Week 24 - pSS
Description: Composite response is defined as the percent of participants with at least 3 of the following at Week 24:
  * Decrease of ≥ 1 point or 15% from baseline in the ESSPRI Total Score
  * Decrease of ≥ 3 points from baseline in ESSDAI score
  * Decrease of ≥ 25% from baseline in ocular staining score, or if normal score at baseline no change to abnormal
  * Increase of ≥ 25% from baseline in stimulated salivary flow
  * Improvement in one or more serological markers (rheumatoid factor (RF), immunoglobulin G protein (IgG), complement C3 or C4, cryoglobulin).
Time Frame: Week 24
Population: All Treated Participants (Prespecified for participants in the pSS cohort only).
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | pSS- Placebo | pSS- Branebrutinib
Number analyzed (Participants) | 4 | 10
Percent of Participants | 25 [0.0 to 67.4] | 10 [0.0 to 28.6]
Statistical Analysis 1: Comparison: pSS- Placebo vs pSS- Branebrutinib; Test type: Superiority — RESPONSE DIFFERENCE (95% CI) VS PLACEBO; Response Difference = -11.9, 95% CI 2-sided [-57.1 to 33.3]
Statistical Analysis 2: Comparison: pSS- Placebo vs pSS- Branebrutinib; Test type: Superiority — ODDS RATIO (95% CI) VS PLACEBO; p = 0.5930, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.40, 95% CI 2-sided [0.02 to 10.02]

5. Primary Outcome: Percent of Participants With ACR50 Response at Week 12 Compared to Baseline - RA
Description: ACR50 response is defined as both improvement of 50% in the number of tender and swollen joints and a 50% improvement in 3 of the following 5 criteria:
  * Subject global assessment (SGA)
  * Physician global assessment (PGA)
  * Functional ability measure
  * Pain visual analog scale (VAS)
  * Erythrocyte sedimentation rate (ESR) or C-reactive protein (CRP).
  Baseline values are defined as the last nonmissing value prior to the first dose of study treatment.
Time Frame: Week 12
Population: All Treated Participants (Prespecified for participants in the RA cohort only).
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | RA- Placebo | RA- Branebrutinib
Number analyzed (Participants) | 21 | 64
Percent of Participants | 33.3 [13.2 to 53.5] | 18.8 [9.2 to 28.3]
Statistical Analysis 1: Comparison: RA- Placebo vs RA- Branebrutinib; Test type: Superiority — RESPONSE DIFFERENCE VS PLACEBO; Response Difference = -14.6, 95% CI 2-sided [-36.9 to 7.7]
Statistical Analysis 2: Comparison: RA- Placebo vs RA- Branebrutinib; Test type: Superiority — ODDS RATIO VS PLACEBO; p = 0.1639, Chi-squared; Odds Ratio (OR) = 0.46, 95% CI 2-sided [0.15 to 1.39]

6. Secondary Outcome: Change From Baseline in DAS28-CRP at Week 12 - RA
Description: The Disease Activity Score-28-C-Reactive Protein (DAS28CRP) is a composite outcome assessment that measures: 1) How many joints in the hands, wrists, elbows, shoulders, and knees are swollen and/or tender over a total of 28, 2) CRP in the blood to measure the degree of inflammation, and 3) SGA of disease activity.
  DAS28-CRP scores range from 1.0 to 9.4, where lower scores indicate less disease activity. The results are combined to produce the DAS28-CRP score, which correlates with the extent of disease activity:
  < 2.6: Disease remission 2.6 - 3.2: Low disease activity 3.2 - 5.1: Moderate disease activity > 5.1: High disease activity
  A negative change from baseline in DAS28-CRP indicates an improvement. Baseline values are defined as the last nonmissing value prior to the first dose of study treatment.
Time Frame: Week 12
Population: All Treated Participants with baseline and week 12 measurements (Prespecified for participants in the RA cohort only).
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | RA- Placebo | RA- Branebrutinib
Number analyzed (Participants) | 19 | 58
Score on a scale | -1.615 (1.19545) | -1.542 (1.0790)
Statistical Analysis 1: Comparison: RA- Placebo; Test type: Equivalence — ADJUSTED MEAN DIFFERENCE WEEK 12; Mean Difference (Final Values) = -1.610, 95% CI 2-sided [-2.110 to -1.110]
Statistical Analysis 2: Comparison: RA- Branebrutinib; Test type: Equivalence — ADJUSTED MEAN DIFFERENCE AT WEEK 12; Mean Difference (Final Values) = -1.567, 95% CI 2-sided [-1.855 to -1.280]
Statistical Analysis 3: Comparison: RA- Placebo vs RA- Branebrutinib; Test type: Superiority — ADJUSTED MEAN DIFFERENCE VS PLACEBO; Mean Difference (Final Values) = 0.043, 95% CI 2-sided [-0.534 to 0.620]

7. Secondary Outcome: Change From Baseline in DAS28-ESR at Week 12 - RA
Description: The Disease Activity Score Erythrocyte Sedimentation Rate - DAS28ESR is a composite outcome assessment that measures:
  1. How many joints in the hands, wrists, elbows, shoulders, and knees are swollen and/or tender over a total of 28
  2. ESR in the blood to measure the degree of inflammation
  3. SGA of disease activity
  DAS28-ESR scores range from 1.0 to 9.4, where lower scores indicate less disease activity. The results are combined to produce the DAS28-ESR score, which correlates with the extent of disease activity:
  < 2.6: Disease remission 2.6 - 3.2: Low disease activity 3.2 - 5.1: Moderate disease activity > 5.1: High disease activity
  A negative change from baseline in DAS28-ESR indicates an improvement. Baseline values are defined as the last nonmissing value prior to the first dose of study treatment.
Time Frame: Week 12
Population: All treated participants with baseline and week 12 measurements (Prespecified for participants in the RA cohort only).
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | RA- Placebo | RA- Branebrutinib
Number analyzed (Participants) | 20 | 58
Score on a scale | -1.758 (1.1932) | -1.670 (1.1487)
Statistical Analysis 1: Comparison: RA- Placebo; Test type: Equivalence — ADJUSTED MEAN DIFFERENCE AT WEEK 12; Mean Difference (Final Values) = -1.741, 95% CI 2-sided [-2.256 to -1.226]
Statistical Analysis 2: Comparison: RA- Branebrutinib; Test type: Equivalence — ADJUSTED MEAN DIFFERENCE AT WEEK 12; Mean Difference (Final Values) = -1.698, 95% CI 2-sided [-1.998 to -1.399]
Statistical Analysis 3: Comparison: RA- Placebo vs RA- Branebrutinib; Test type: Superiority — ADJUSTED MEAN DIFFERENCE VS PLACEBO; Mean Difference (Final Values) = 0.043, 95% CI 2-sided [-0.553 to 0.639]

8. Secondary Outcome: Change From Baseline in SDAI at Week 12- RA
Description: The Simplified Disease Activity Index (SDAI) is the sum of the tender joint score (range 0 to 28), the swollen joint score (range 0 to 28), the subject global assessment (SGA) of disease activity (range 0 to 10 in increments of 0.5), the PGA of disease activity (range 0 to 10 in increments of 0.5), and C-reactive protein (CRP) test result. Baseline values are defined as the last nonmissing value prior to the first dose of study treatment. A SDAI score ranges from 0 (disease remission) to 86 (high disease activity).
Time Frame: Week 12
Population: All treated participants with baseline and week 12 measurements (Prespecified for participants in the RA cohort only).
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | RA- Placebo | RA- Branebrutinib
Number analyzed (Participants) | 19 | 58
Score on a scale | -19.430 (12.5890) | -18.303 (11.5793)
Statistical Analysis 1: Comparison: RA- Placebo; Test type: Equivalence — ADJUSTED MEAN DIFFERENCE AT WEEK 12; Mean Difference (Final Values) = -19.495, 95% CI 2-sided [-24.861 to -14.128]
Statistical Analysis 2: Comparison: RA- Branebrutinib; Test type: Equivalence — ADJUSTED MEAN DIFFERENCE AT WEEK 12; Mean Difference (Final Values) = -18.767, 95% CI 2-sided [-21.848 to -15.686]
Statistical Analysis 3: Comparison: RA- Placebo vs RA- Branebrutinib; Test type: Superiority — ADJUSTED MEAN DIFFERENCE VS PLACEBO; Mean Difference (Final Values) = 0.728, 95% CI 2-sided [-5.463 to 6.919]

9. Secondary Outcome: Change From Baseline in CDAI at Week 12 - RA
Description: The Clinical Disease Activity Index (CDAI) is the sum of the tender joint score (range 0 to 28), the swollen joint score (range 0 to 28), the SGA of disease activity (range 0 to 10 in increments of 0.5), and the PGA of disease activity (range 0 to 10 in increments of 0.5). Baseline values are defined as the last nonmissing value prior to the first dose of study treatment. A CDAI score ranges from 0 to 76.
  The interpretation of CDAI is as follows:
  0.0 - 2.8: Disease remission 2.9 - 10.0: Low disease activity (LDA) 10.1 - 22.0: Moderate disease activity 22.1 - 76.0: High disease activity
Time Frame: Week 12
Population: All treated participants with baseline and week 12 measurements (Prespecified for participants in the RA cohort only).
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | RA- Placebo | RA- Branebrutinib
Number analyzed (Participants) | 20 | 58
Score on a scale | -19.4 (12.07) | -18.0 (11.01)
Statistical Analysis 1: Comparison: RA- Placebo; Test type: Equivalence — ADJUSTED MEAN AT DIFFERENCE WEEK 12; Mean Difference (Final Values) = -19.2, 95% CI 2-sided [-24.3 to -14.1]
Statistical Analysis 2: Comparison: RA- Branebrutinib; Test type: Equivalence — ADJUSTED MEAN AT DIFFERENCE WEEK 12; Mean Difference (Final Values) = -18.5, 95% CI 2-sided [-21.4 to -15.5]
Statistical Analysis 3: Comparison: RA- Placebo vs RA- Branebrutinib; Test type: Superiority — ADJUSTED MEAN DIFFERENCE VS PLACEBO; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-5.2 to 6.6]

10. Secondary Outcome: Percent of Participants With ACR20 Response Compared to Baseline at Week 12 - RA
Description: ACR20 defined as both improvement of 20% in the number of tender and swollen joints and a 20% improvement in 3 of the following 5 criteria:
  * Subject global assessment (SGA)
  * Physician global assessment (PGA)
  * Functional ability measure
  * Pain visual analog scale (VAS)
  * Erythrocyte sedimentation rate (ESR) or C-reactive protein (CRP).
  Baseline values are defined as the last nonmissing value prior to the first dose of study treatment.
Time Frame: Week 12
Population: All Treated Participants (Prespecified for participants in the RA cohort only).
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | RA- Placebo | RA- Branebrutinib
Number analyzed (Participants) | 21 | 64
Percent of Participants | 61.9 [41.1 to 82.7] | 57.8 [45.7 to 69.9]
Statistical Analysis 1: Comparison: RA- Placebo vs RA- Branebrutinib; Test type: Superiority — RESPONSE DIFFERENCE VS PLACEBO; Response Difference = -4.1, 95% CI 2-sided [-28.1 to 19.9]
Statistical Analysis 2: Comparison: RA- Placebo vs RA- Branebrutinib; Test type: Superiority — ODDS RATIO VS PLACEBO; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.31 to 2.32]

11. Secondary Outcome: Percent of Participants With ACR70 Response Compared to Baseline at Week 12 - RA
Description: ACR70 is defined as both improvement of 70% in the number of tender and swollen joints and a 70% improvement in 3 of the following 5 criteria:
  * Subject global assessment (SGA)
  * Physician global assessment (PGA)
  * Functional ability measure
  * Pain visual analog scale (VAS)
  * Erythrocyte sedimentation rate (ESR) or C-reactive protein (CRP).
  Baseline values are defined as the last nonmissing value prior to the first dose of study treatment.
Time Frame: Week 12
Population: All Treated Participants (Prespecified for participants in the RA cohort only).
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | RA- Placebo | RA- Branebrutinib
Number analyzed (Participants) | 21 | 64
Percent of Participants | 14.3 [0.0 to 29.3] | 7.8 [1.2 to 14.4]
Statistical Analysis 1: Comparison: RA- Placebo vs RA- Branebrutinib; Test type: Superiority — RESPONSE DIFFERENCE VS PLACEBO; Response Difference = -6.5, 95% CI 2-sided [-22.8 to 9.9]
Statistical Analysis 2: Comparison: RA- Placebo vs RA- Branebrutinib; Test type: Superiority — ODDS RATIO VS PLACEBO; Odds Ratio (OR) = 0.51, 95% CI 2-sided [0.11 to 2.34]

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from participants first dose to their study completion (up to approximately 32 weeks) SAEs and Other AEs were assessed from first dose to 30 days following last dose (up to approximately 30 weeks)
Description: TEAEs are defined as AEs that occur after the participant received first dose of study treatment or if a preexisting condition worsens in severity or becomes serious after receiving the first dose of study treatment up to 30 days after the last dose of study treatment.
Groups:
- RA- Branebrutinib: Participants with rheumatoid arthritis (RA) receive branebrutinib 9mg once daily (QD) during a 12-week double-blind placebo-controlled treatment period.
- RA Abatacept: Participants with rheumatoid arthritis (RA) receive 12 weeks of treatment with open-label abatacept after the 12-week double-blind placebo-controlled treatment period.
Arm/Group | SLE- Placebo | SLE- Branebrutinib | pSS- Placebo | pSS- Branebrutinib | RA- Placebo | RA- Branebrutinib | RA Abatacept
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/15 | 0/4 | 0/10 | 0/21 | 0/64 | 0/81
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/15 | 0/4 | 0/10 | 0/21 | 0/64 | 0/81
Other Adverse Events (participants affected / at risk) | 4/5 | 14/15 | 4/4 | 8/10 | 6/21 | 13/64 | 5/81
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SLE- Placebo (N=5) | SLE- Branebrutinib (N=15) | pSS- Placebo (N=4) | pSS- Branebrutinib (N=10) | RA- Placebo (N=21) | RA- Branebrutinib (N=64) | RA Abatacept (N=81)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 5 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2 | 3 | 2 | 1 | 1 | 1
Otitis media acute (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 3 | 0 | 1 | 0 | 0 | 1
Animal scratch (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Face injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 1 | 0
Gastric pH decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 1 | 1 | 1 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 0
Stress (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT04186871/Prot_SAP_000.pdf